CLINICAL TRIAL: NCT06059586
Title: Pre-Rehabilitation for Female Patients Undergoing Pelvic Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Namita Agrawal, Assistant Professor of Radiation Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO-IUSCCC-0772
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Dyspareunia; Pelvic Pain; Sexual Dysfunction; Radiation Toxicity
Keywords: vaginal dilator; pelvic health physical therapy
MeSH Terms: conditions — Dyspareunia; Pelvic Pain; Sexual Dysfunction, Physiological; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pelvic health Assessment and Intervention (Experimental)
  Interventions: Behavioral: Pelvic health therapy; Device: Dilator feasability

INTERVENTIONS:
Behavioral: Pelvic health therapy — Female Sexual Function Index (FSFI) and VAS Pain Scale Questionnaires, Physical Therapy Evaluation including Pelvic Floor Muscle Examination, Dilator Education
Device: Dilator feasability — Patient Adherence to Vaginal Dilation Questionnaire

SUMMARY:
The purpose of this study is to examine the feasibility of adding pre-rehabilitation pelvic health physical therapy to standard of care radiation therapy treatment plan for female patients who have been diagnosed with cervical, vaginal, vulvar, uterine, or anal cancer and are a candidate for curative pelvic radiation with external beam. Participants will receive education on using a vaginal dilator for use during treatment and complete questionnaires looking at pain and sexual function.

DETAILED DESCRIPTION:
Because of the increasing survivorship rate, there is a need for research addressing the post-treatment side effects of pelvic pain and dyspareunia, due to the significant impact these side effects have on patients' quality of life. Current best practice from trained pelvic health physical therapists for addressing dyspareunia and pelvic pain due to vaginal stenosis after radiation therapy, is vaginal dilation. Vaginal dilators are cone shaped durable medical equipment that are inserted into the vagina with lubricant, to assist in patency of the vaginal canal and stretching of the pelvic floor muscles.

The primary objective of this pilot clinical trial is to assess the feasibility of implementing a collaborative, coordinated, and multidisciplinary initiative between radiation oncology and pelvic health physical therapy to answer the following questions: 1) What are the barriers and facilitators to the implementation of a pre-rehabilitation service for gynecological and female anal cancer patients undergoing pelvic radiation and 2) What is the potential clinical value of adding pre-rehabilitative pelvic health services, with an emphasis on vaginal dilator education and use, to the gynecological and female anal cancer radiation setting, in collaboration with radiation oncology staff, as a means of reducing pelvic pain and dyspareunia?

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. ≥ 18 years old at the time of informed consent
3. Ability to provide written informed consent and HIPAA authorization
4. Primary diagnosis of cervical, vaginal, vulvar, uterine, or anal cancer
5. Candidate for curative pelvic radiation with external beam, with or without brachytherapy, per radiation oncologist's discretion

Notes:

* Can have prior and/or current modalities of treatment to address diagnosis including surgery and chemotherapy
* Can receive radiation at any facility provided patient is able to perform Physical Therapy visits at IUH North/Schwarz Cancer Center

Exclusion Criteria:

1. Major medical illnesses or psychiatric impairments, which in the investigator's opinion will prevent administration or completion of the protocol therapy and/or interfere with follow-up.
2. Not a candidate for curative radiation therapy per radiation oncologist's discretion
3. Prior radiation therapy to the pelvis
4. Women who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasability of implementation of pre-rehabilitation to radiotherapy | Baseline
  Recording the number of eligible patients for protocol that decline enrollment. The reason(s) for forgoing protocol intervention will be documented.
Feasability of implementation of pre-rehabilitation to radiotherapy | Baseline
  The number of eligible patients that were not identified for protocol enrollment will be recorded and potential gaps in the screening process will be analyzed.
Feasability of implementation of pre-rehabilitation to radiotherapy | Baseline
  The number of eligible patients identified, but not screened, for eligibility or not consented if eligible will be recorded.
Feasability of implementation of pre-rehabilitation to radiotherapy | Baseline
  The duration of time from initial clinical presentation to being offered information of clinical study will be recorded.
Feasability of implementation of pre-rehabilitation to radiotherapy | Baseline to 6 weeks
  The duration of time from enrollment on clinical study to being seen by physical therapy will be recorded.
Feasability of implementation of pre-rehabilitation to radiotherapy | Baseline to 4 months
  The number of Female Sexual Function Index questionnaires will be recorded as completed, incomplete or not attempted. Reasons for submitting incomplete questionnaires or not submitting a questionnaire will be recorded.

SECONDARY OUTCOMES:
Average score on the Visual Pain Rating Scale. | Immediately upon radiation completion, 4 weeks, 6 weeks, 8 weeks, 12 weeks, and 16 weeks post radiation
  Visual Analogue Pain Rating Scale 0-10
Evaluate female sexual function based on questionnaire responses | Immediately upon radiation completion, 4 weeks, 6 weeks, 8 weeks, 12 weeks, and 16 weeks post radiation
  Female Sexual Function Index questionnaires (Likert scale)
Percentage of adherence to dilator use | Immediately upon radiation completion, 4 weeks, 6 weeks, 8 weeks, 12 weeks, and 16 weeks post radiation
  Self-reported dilator adherence

CONTACTS AND LOCATIONS:
Overall Officials: Namita Agrawal, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Health West, Avon, Indiana
  - IU Health Schwarz Cancer Center, Carmel, Indiana